CLINICAL TRIAL: NCT06216002
Title: Incidence of Residual Neuromuscular Blockade in Patients With Frailty Undergoing Gynecologic Cancer Surgery
Brief Title: Incidence of Residual Neuromuscular Blockade in Fraility in OncoGynae Surgery
Acronym: FIGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 599/2566(IRB3)
Record Dates: First submitted 2023-11-13; First posted 2024-01-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Frailty; Neuromuscular Blockade; General Anesthetic Drug Adverse Reaction; Gynecologic Cancer; Surgical Complication
Keywords: neuromuscular blocking agents; frailty; gynecologic oncology; surgery; anesthetic complications
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Train of four nerve stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TOF nerve stimulation (Experimental): Patient receive TOF nerve stimulation in recovery room after surgery
  Interventions: Diagnostic Test: Train of four nerve stimulator

INTERVENTIONS:
Diagnostic Test: Train of four nerve stimulator — Patient receive nerve stimulation by TOF-scan equipment at recovery room after surgery.

SUMMARY:
Frailty among patients undergoing surgery is strongly associated with an elevated risk of adverse perioperative outcomes, heightened incidence of postoperative complications, increased mortality rates, and prolonged hospital length of stay. Our focus centers on investigating the frailty index in the context of complications experienced by patients undergoing oncologic gynecology surgery. The principal objective of this research is to elucidate the extent to which residual neuromuscular blocking agents are linked to frailty.

DETAILED DESCRIPTION:
Among patients undergoing oncologic gynecological procedures, such as those for vulvar cancer, endometrial cancer, and ovarian cancer, the incidence of frailty has been observed to range from 14% to 45%. Frailty directly influences the metabolism of anesthetic agents and intraoperative management. Furthermore, the prevalence of residual neuromuscular blocking agents following surgery can be as high as 26% to 53%. No prior research has investigated the correlation between residual muscle relaxants and frailty in gynecologic oncology patients. This study is designed to assess the prevalence of residual muscle relaxants in these patients with frailty. Additionally, data on the incidence of frailty and its impact on postoperative outcomes and prognosis in patients undergoing gynecologic oncology surgery will be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

* Age >,= 18 years
* Patients undergoing elective gynecologic-oncology surgery

Exclusion Criteria:

* Unable to communicate Thai
* Unable to understand the questionnaire
* Preexisting neuromuscular disease
* Preexisting disease involved wrist that may affect the nerve stimulator examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of residual neuromuscular blockade | 0-30 minute after surgery
  Incidence of residual neuromuscular blockade with the relation of frailty after gynecologic oncology surgery
Incidence of frailty | 0 - 24 hours preoperative
  Incidence of frailty in patients undergoing gynecologic oncology surgery

SECONDARY OUTCOMES:
Anesthetic technique used | Throughout Intraoperative period, an average 3-5 hours
  Anesthetic technique used in patients undergoing gynecologic oncology surgery
Rate of blood transfusion | Throughout Intraoperative period, an average 3-5 hours to 24 hours postoperative
  Quantity of units blood transfusion
Rate of vasopressor usage | Throughout Intraoperative period, an average 3-5 hours to 24 hours postoperative
  Rate of vasopressor usage eg. ephedrine, norepinephrine
Length of hospital stay | Through study completion, an average of 1 year, an average 3 - 5 days
  Total number of days of hospital stay
Rate of intensive care unit admission | 0 - 24 hours postoperative
  Number of patients who require intensive care unit admission after surgery
Rate of re-intubation | 0 - 24 hours postoperative
  Number of patients who require re-intubation
Rate of postoperative mechanical ventilation | 0 - 24 hours postoperative
  Number of patients who require mechanical ventilation postoperative
Rate of postoperative pulmonary complications | 3 days after operation
  Number of patients who have postoperative pulmonary complications eg. prolonged intubation, atelectasis, pneumonia etc.
Mortality rate | 30 days after operation
  Number of patients who died after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Study Director — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University; Jitsupa Nithiuthai, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No